CLINICAL TRIAL: NCT01285856
Title: Hair Testing to Assess Consumption of Illicit Psychotropic Agents and Alcohol by Patients Treated With High-dose Buprenorphine and Methadone. Search for a Pharmacogenetic Contribution to Low Efficacy of Substitution Medications
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Assistance Publique Hopitaux De Marseille (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None
Other Study IDs: 2010-A00256-33; 2010-A00256-33 (Other: DRC)
Record Dates: First submitted 2010-07-29; First posted 2011-01-28 (Estimated); Last update posted 2014-08-29 (Estimated); Status verified 2014-08

CONDITIONS: Substance Abuse
Keywords: patients; illicit consumption of psychotropic agents and alcohol; buprenorphine; methadone
MeSH Terms: conditions — Substance-Related Disorders

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- buprenorphine (Active Comparator): populations of patients treated with HDB will be recruited during consultations at a center for addiction treatment. One hundred and ten patients will be included. Written informed consent will be obtained from each patient. Anonymity will be respected at inclusion and throughout. Using a sample of hair, testing for and measurement of the principal drugs (opiates, cannabis, cocaine, amphetamines) and the specific marker of ethanol consumption, ethyl glucuronide, will be performed by chromatographic techniques (high-performance liquid chromatography and gas phase chromatography) together with detection by mass or tandem mass spectrometry. Treatment efficacy will also be assessed using Handelsman's subjective and objective opiate withdrawal scales. Lastly, polymorphisms of the metabolic enzymes of methadone and HDB will be sought by real-time PCR in a saliva sample, a method which gives similar results without the need for venous blood sampling.
  Interventions: Other: hair and saliva samples
- methadone (Active Comparator): populations of patients treated with methadone will be recruited during consultations at a center for addiction treatment. One hundred and ten patients will be included. Written informed consent will be obtained from each patient. Anonymity will be respected at inclusion and throughout. Using a sample of hair, testing for and measurement of the principal drugs (opiates, cannabis, cocaine, amphetamines) and the specific marker of ethanol consumption, ethyl glucuronide, will be performed by chromatographic techniques (high-performance liquid chromatography and gas phase chromatography) together with detection by mass or tandem mass spectrometry. Treatment efficacy will also be assessed using Handelsman's subjective and objective opiate withdrawal scales. Lastly, polymorphisms of the metabolic enzymes of methadone and HDB will be sought by real-time PCR in a saliva sample, a method which gives similar results without the need for venous blood sampling.
  Interventions: Other: hair and saliva samples

INTERVENTIONS:
Other: hair and saliva samples — Using a sample of hair, testing for and measurement of the principal drugs (opiates, cannabis, cocaine, amphetamines) and the specific marker of ethanol consumption, ethyl glucuronide, will be performed by chromatographic techniques (high-performance liquid chromatography and gas phase chromatography) together with detection by mass or tandem mass spectrometry. This non-invasive sampling is more informative than blood tests, as it gives a retrospective profile of an individual's consumption over several months.
  Saliva sample, a method which gives similar results without the need for venous blood sampling.

SUMMARY:
Justification and aims of the study: The principal aim of use of opiate substitutes such as methadone or high-dose buprenorphine (HDB) is to reduce the need or the desire to consume the opiate to which the patient is addicted. Adjustment of the initial dose and regular re-evaluation of the efficacy of treatment are key elements in the success of such management. While too high a dose can be responsible for side effects leading to abandonment of treatment, too low a dose can induce the reappearance or even the reinforcing of parallel consumption of other psychoactive substances, in particular cocaine, alcohol and cannabis. The principal aim of this project is to determine the course of parallel consumption in patients who have been receiving a maintenance dose of methadone or HDB for at least two months, by analysis of a sample of hair, a biological matrix which is innovative for this type of study. Hair testing establishes a retrospective profile of consumption. The secondary aims of this project are (i) to validate the French versions of Handelsman's subjective and objective opiate withdrawal scales and to seek a possible correlation between high scores on these scales and the presence of parallel consumption, and (ii) to seek an association between polyconsumption and common functional polymorphisms of metabolic enzymes of methadone and HDB.

Expected results: Hair testing, which has the particular advantage of a long detection window so that samples need only be taken at intervals, could improve the biological monitoring of patients on substitutive treatment.

Validation of the French version of Handelsman's scales of objective and subjective signs of opiate withdrawal and search for any correlation with parallel consumption will enable these scales to be used in daily practice for clinical surveillance of patients on substitutive treatment.

If a polymorphism of a metabolic enzyme of one or other of these molecules is detected, rapid genotyping of a simple saliva sample will be valuable in guiding the choice of medication when deciding on a treatment strategy

DETAILED DESCRIPTION:
Methodology: The two populations of patients, one treated with methadone, the other with HDB, will be recruited in accordance with the ethical principles of the declaration of Helsinki, during consultations at a center for addiction treatment. One hundred and ten patients will be included in each of the two populations. Written informed consent will be obtained from each patient. Anonymity will be respected at inclusion and throughout. Using a sample of hair, testing for and measurement of the principal drugs (opiates, cannabis, cocaine, amphetamines) and the specific marker of ethanol consumption, ethyl glucuronide, will be performed by chromatographic techniques (high-performance liquid chromatography and gas phase chromatography) together with detection by mass or tandem mass spectrometry. This non-invasive sampling is more informative than blood tests, as it gives a retrospective profile of an individual's consumption over several months. Treatment efficacy will also be assessed using Handelsman's subjective and objective opiate withdrawal scales. Lastly, polymorphisms of the metabolic enzymes of methadone and HDB will be sought by real-time PCR in a saliva sample, a method which gives similar results without the need for venous blood sampling.

ELIGIBILITY:
Inclusion Criteria:

* subjects followed for opiates substitute treatment
* patients treated by HDB or methadone for at least two months
* length of hair superior to 2 centimeters

Exclusion Criteria:

* patients treated by HDB or methadone for less than two months
* Patients with clinical signs of intolerance or opioid overdose
* opioid treatments
* neurological or psychiatric disease
* hepatic disease
* pregnancy
* patients in prison

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 220 (Estimated)
Dates: Start 2010-08; Primary Completion 2015-08 (Estimated); Study Completion 2015-08 (Estimated)

PRIMARY OUTCOMES:
Hair ANALYSIS | 36 months
  Hair testing which has the particular advantage of a long detection window so that samples need only be taken at intervals

SECONDARY OUTCOMES:
Validation of the French version of Handelsman's scales | 36 months
  Validation of the French version of Handelsman's scales of objective and subjective signs of opiate withdrawal and search for any correlation with parallel consumption will enable these scales to be used in daily practice for clinical surveillance of patients on substitutive treatment.
polymorphism of a metabolic enzyme | 36 months
  If a polymorphism of a metabolic enzyme of one or other of these molecules is detected, rapid genotyping of a simple saliva sample will be valuable in guiding the choice of medication when deciding on a treatment strategy.

CONTACTS AND LOCATIONS:
Overall Officials: Anne-Laure Pelissier-Alicot, Principal Investigator — APHM
Locations (1):
- APHM, Marseille, France